CLINICAL TRIAL: NCT03364972
Title: A Randomised, Controlled Study to Compare Visual Performance, Refractive Outcome, Forward Light Scatter, Patient Satisfaction and Objective Measurement of Glistenings Following Insertion of Two Monofocal, Aspheric, Hydrophobic Acrylic Intraocular Lenses: the Alcon CLAREON® and the Abbott Medical Optics PCB00 Lenses
Brief Title: A Study Comparing Two Monofocal, Aspheric, Hydrophobic Acrylic Intraocular Lenses: the Alcon CLAREON® and the Abbott Medical Optics PCB00
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 232017
Record Dates: First submitted 2017-11-21; First posted 2017-12-07 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Cataract Extraction; Phacoemulsification; Glistenings; Intraocular Lens Implant; Hydrophobic Acrylic; Cataract Surgery; Light Scatter; Patient Satisfaction; Patient Related Outcome Measures
Keywords: cataract; cataract extraction; interocular lens implant; glistenings; phacoemulsification; hydrophobic acrylic; light scatter; patient related outcome measures
MeSH Terms: conditions — Patient Satisfaction; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intraocular lens implant (Experimental): 'Alcon Clareon' : New monofocal, hydrophobic acrylic intraocular lens implant
  Interventions: Device: Cataract surgery
- Standard intraocular lens implant (Active Comparator): Abbott Tecnis PCB00- Standard monofocal,hydrophobic acrylic intraocular lens implant
  Interventions: Device: Cataract surgery

INTERVENTIONS:
Device: Cataract surgery — Conventional small-incision phacoemulsification cataract surgery with insertion of intraocular lens implant

SUMMARY:
This is a bilateral randomised controlled study to compare visual performance, refractive outcome, forward light scatter, patient satisfaction and objective measurement of glistenings following insertion of two monofocal, aspheric, hydrophobic acrylic intraocular lenses (IOLs). A new product is compared with an established one.

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataracts
* good visual potential
* ability to understand informed consent and objectives of the trial
* not-pregnant
* not breast feeding
* no previous eye surgery
* corneal astigmatism less than 1 diopter in both eyes

Exclusion Criteria:

* age-related macula degeneration
* glaucoma
* previous retinal vascular disorders
* previous retinal detachment or tear
* any neuro-ophthalmological condition
* any inherited retinal disorder or pathology
* previous strabismus surgery or record of amblyopia
* previous transient ischaemic attacks, cerebrovascular events or other vaso-occlusive disease
* already enrolled in another study
* Exclusion criteria relate to clinical contraindications for Femtosecond Laser Assisted Cataract Surgery, such as:

  * Significant corneal opacities
  * Small pupils following pharmacological dilatation
  * Patients unable to lie sufficiently flat so as to be positioned underneath the laser machine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 13 months
  As measured by conventional LogMAR visual acuity charts

SECONDARY OUTCOMES:
Incidence of intraocular lens glistenings | 13 months
  Incidence of presence of intraocular lens glistenings in each study arm
Severity of intraocular lens glistenings | 13 months
  Number of vacuoles per square millimetre
Refraction (i.e. glasses prescription) | 13 months
  In conventional sphere/cylinder dioptre scales: total range -40 to +40, in 0.25 steps. Higher values represent worse outcome. Values closer to 0 (zero) represent better outcome

OTHER OUTCOMES:
Forward light scatter | 13 months
  Intraocular (forward) light scatter is measured with a specifically devised computerised vision test. It is represented by straylight parameter, Log(s), on a logarithmic scale from 0 to 1.5. The lower the value (i.e. closer to 0), the better the outcome.
Contrast sensitivity | 13 months
  Visual acuity (LogMAR scale: total range -0.2 to 1.0 in 0.02 steps) measured at different contrasts with a computerized contrast sensitivity chart. Negative values, or values closer to 0, represent better outcome.
Patient satisfaction | 13 months
  Validated patient satisfaction questionnaire. We use specially designed and validated conversion tables to convert raw scores from questionnaires to Rasch calibrated measures.
Self-reported health | 13 months
  Validated self-reported health questionnaire. We use a vertical Visual Analogue Scale (VAS) to record patients' self-reported health on a scale from 0-100 (values closer or equal to 100 represent better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- St Thomas' Hospital NHS Trust, London, United Kingdom